CLINICAL TRIAL: NCT02088229
Title: Relating Retinal Structural and Functional Parameters to Visual Acuity in Eyes Undergoing Treatment for Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Grant Comer, Edward T and Ellen K Dryer Career Development Professor of Ophthalmology and Visual Sciences and Assistant Professor of Ophthalmology and Visual Sciences, Medical School, University of Michigan
Other Study IDs: HUM00064483
Record Dates: First submitted 2014-03-07; First posted 2014-03-14 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This longitudinal interventional case series will utilize the patients at the University of Michigan W.K. Kellogg Eye Center scheduled to begin treatment for diabetic macular edema. Baseline measures will be taken which include structural assessments such as circulatory capacity utilizing fluorescein angiography, in addition to retinal layer integrity and thickness using high resolution optical coherence tomography. Also, functional assessments such as visual acuity, contrast sensitivity, photostress recovery, dark adaptation, perimetry, and cellular fluorescence will be tested. Adverse events will be recorded and compared with historical controls to ensure that currently accepted interventions are safe. Finally, potential confounding variables for DME including those related to the eye, systemic factors, and patient demographics will be recorded to assess the influence of these variables on treatment response.

The primary objective is to develop hypotheses that might better explain the retinal structural (anatomical) and/or functional (physiological) mechanisms of visual impairment in eyes receiving treatment for diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Males and females age ≥ 18 years
* DME involving the central fovea (≥325 micrometers central subfield thickness on Spectralis SD-OCT)
* Scheduled to undergo treatment of DME with intravitreal bevacizumab or ranibizumab
* Willing to sign informed consent, comply with study protocol requirements, and undergo at least 2.5 hours of testing per visit;

Exclusion Criteria:

* Lens opacity ≥ grade 3 ARLNS on standard photographs
* Incisional ophthalmic surgery of any kind within 4 months of study enrollment
* Treatment for DME within the past 4 months
* Active proliferative diabetic retinopathy
* History of vitrectomy
* Glaucoma
* Uncontrolled hypertension (≥ 180 systolic or ≥ 110 diastolic on two successive measures)
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception throughout the study
* Females who are pregnant, lactating or breastfeeding at time of enrollment
* Subjects with a history of a serious hypersensitivity reaction to treatment or components of the study assessment
* History of any radiation in or around the eyes
* History of visually significant non-diabetic retinopathy or choroidopathy (e.g. age-related macular degeneration, polypoidal choroidal vasculopathy, central serous retinopathy, retinal vein occlusion, sickle cell retinopathy)
* History of optic neuropathy
* Neurological conditions that can impair vision (e.g. Parkinson's disease, multiple sclerosis, Alzheimer's disease)
* Liver disease (e.g. cirrhosis, hepatitis)
* History of small bowel surgery
* Anticipated need for intravitreal triamcinolone injections
* Dilated pupil diameter less than 6 millimeters
* High myopia (refractive error spherical equivalent ≥ -6 diopters)
* Currently being treated for cancer or any disease likely to adversely affect participation in a 2 year trial
* Participation in any interventional clinical study requiring IRB approval within 3 months of enrollment
* Any findings deemed unacceptable by the Principal Investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing treatment for diabetic macular edema at the University of Michigan W.K. Kellogg Eye Center.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Dark adaptation (AdaptRx) | 12 Months
  Rod intercept (minutes)

SECONDARY OUTCOMES:
Optical coherence tomography | 12 Months
  Thickness of nerve fiber layer and ganglion cell layer, volume of intraretinal cysts, volume of subretinal fluid, central subfield thickness, thickness of choroid (enhanced depth imaging), status of vitreoretinal interface, presence of epiretinal membrane, status of inner segment/outer segment junction

OTHER OUTCOMES:
Fluorescein angiography | 12 months
  Fluorescein transit time, foveal avascular zone (FAZ) greatest linear dimension, FAZ area, presence of perifoveal capillary loss, area of dye leakage, and microaneurysm density
Lipofuscin fundus autofluorescence | 12 Months
  Index of retinal autofluorescence
Color photographs | 12 Months
  Diabetic Retinopathy Disease Severity Scale
Frequency Doubling Threshold visual field | 12 Months
  Mean deviation, pattern standard deviation
Contrast sensitivity | 12 Months
  Log contrast sensitivity
Photostress test | 12 Months
Flavoprotein fluorescence | 12 Months
  Index of metabolic fluorescence, average intensity (grey scale unit (gsu)), average curve width (GSU), heterogeneity score

CONTACTS AND LOCATIONS:
Overall Officials: Grant Comer, M.D., Principal Investigator — University of Michigan
Locations (1):
- Kellogg Eye Center, Ann Arbor, Michigan, United States